CLINICAL TRIAL: NCT07002593
Title: Comparative Efficacy of Myofascial Release Versus Stretching Combined With High-Powered Pulsed Therapeutic Ultrasound in Athletes With Active Trapezius Trigger Points: A Randomized Comparative Trial
Brief Title: Myofascial Release vs. Stretching With Ultrasound for Trapezius Trigger Points in Athletes: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, AMIR IQBAL, Principle Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RRC-2022-07
Record Dates: First submitted 2025-05-25; First posted 2025-06-03 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Active Trapezius Trigger Point Pain
Keywords: Myofascial Pain Syndromes; Ultrasonic Therapy; Athletes; Trigger Points; Range of Motion
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Myofascial Release Therapy; Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MFR Group (Experimental): MFR Group received a 10-minute manual myofascial release (MFR) technique followed by a 5-minute session of high-powered pulsed therapeutic ultrasound (HPPT-US). It was performed three times per week for two weeks.
  Interventions: Other: Myofascial release (MFR); Other: High-powered pulsed therapeutic ultrasound (HPPT-US)
- Stretching Group (Active Comparator): Stretching Group received three 30-second static stretches for the upper trapezius, involving neck side flexion with contralateral rotation, followed by a 5-minute session of HPPT ultrasound. It was performed three times per week for two weeks.
  Interventions: Other: Muscle Stretching; Other: High-powered pulsed therapeutic ultrasound (HPPT-US)

INTERVENTIONS:
Other: Myofascial release (MFR) — A 10-minute manual myofascial release (MFR) technique targeting active upper trapezius trigger points (MTrPs), applying sustained pressure until tissue release was achieved.
  Arms: MFR Group
Other: Muscle Stretching — Three 30-second static muscle stretches were performed for the upper trapezius by placing neck side flexion with contralateral rotation.
  Arms: Stretching Group
Other: High-powered pulsed therapeutic ultrasound (HPPT-US) — A 5-minute high-powered pulsed therapeutic ultrasound (HPPT) was delivered subcutaneously with specific parameters of 1.5 W/cm², 1 MHz, and pulsed mode.

SUMMARY:
This study aimed to compare the efficacy of MFR plus HPPT-US versus stretching plus HPPT-US on pain intensity, cervical range of motion (ROM), muscle length (ML), and neck disability in athletes with active upper trapezius MTrPs. Methods: A randomized clinical trial was conducted on 60 male athletes diagnosed with active upper trapezius MTrPs. Participants were randomly assigned to Group A (MFR + HPPT-US) or Group B (stretching + HPPT-US). Interventions were administered over two weeks. Outcome measures including Visual Analog Scale (VAS), ROM, ML, and Neck Disability Index (NDI) were recorded at baseline, week 1, week 2, and one-week follow-up. Between-group comparisons were analyzed using independent t-tests, and effect sizes were calculated using Cohen's d. For all statistical analyses, the level of significance alpha was set at 95% (p < .05).

DETAILED DESCRIPTION:
Neck pain caused by active myofascial trigger points (MTrPs) in the upper trapezius is a significant concern for athletes, often leading to decreased mobility, persistent discomfort, and compromised performance. Research indicates that these hyperirritable muscle knots contribute not only to localized pain but also to referred discomfort and motor dysfunction, creating a cycle of chronic impairment (Simons et al., 1999). The underlying mechanisms involve both peripheral factors-such as inflammation and nerve sensitization-and central nervous system adaptations that amplify pain perception (Fernández-de-las-Peñas & Dommerholt, 2018). The resulting limitations extend beyond physical symptoms, affecting training consistency, competition readiness, and long-term athletic careers (Hoy et al., 2014; Elabd et al., 2024).

Athletic Susceptibility to MTrPs Athletes engaged in repetitive or high-load movements are particularly vulnerable to upper trapezius MTrPs. Sports like swimming, tennis, and weightlifting, which demand sustained shoulder and neck exertion, frequently lead to muscle overuse and microtrauma (Page, 2012). Similarly, disciplines requiring prolonged static postures, such as cycling or wrestling, place continuous strain on the cervical musculature, increasing the likelihood of trigger point development (Wiewelhove et al., 2019). Without effective intervention, these issues can evolve into chronic pain syndromes, further hindering athletic output.

Current Therapeutic Approaches

Management of MTrPs typically involves a multimodal approach, including:

Stretching Techniques - Both static and dynamic methods aim to restore muscle pliability and enhance joint mobility (Behm et al., 2021).

Myofascial Release (MFR) - Hands-on or instrument-assisted techniques target fascial tightness, improving tissue flexibility and reducing stiffness (Cheatham et al., 2015).

High-Power-Pain-Threshold (HPPT) Ultrasound - This modality may accelerate healing by increasing blood circulation and breaking down adhesions within affected muscle fibers (Watson, 2008).

While these treatments are commonly used, the optimal combination remains unclear. Some studies suggest that integrating MFR with HPPT ultrasound could offer synergistic benefits by simultaneously addressing soft tissue restrictions and enhancing cellular repair (Robertson et al., 2016). However, direct comparisons between MFR-based and stretching-focused approaches, particularly in athletes, are lacking.

Study Objective and Expected Outcomes This investigation seeks to determine whether MFR combined with HPPT ultrasound outperforms stretching combined with HPPT ultrasound in alleviating neck pain and restoring function in athletes with active MTrPs. Key measures include pain reduction, cervical mobility, strength recovery, and sport-specific functionality.

Given MFR's ability to directly manipulate fascial restrictions and improve neuromuscular coordination, it is anticipated that this approach will yield greater clinical benefits than stretching alone. The findings could influence rehabilitation protocols, offering athletes more effective strategies to manage myofascial pain and expedite return to peak performance.

Broader Implications By clarifying the most effective treatment combination, this research has the potential to refine sports medicine practices, reducing reliance on temporary pain relief and promoting long-term musculoskeletal health. Enhanced intervention strategies may also decrease the economic burden associated with prolonged athlete downtime, benefiting both individuals and sports organizations.

Ultimately, this study aims to advance evidence-based care for myofascial pain, ensuring athletes receive targeted, efficient therapies that support sustained competitive success.

ELIGIBILITY:
Inclusion Criteria:

* Male athletes
* Aged between 20-40 years
* Active MTrPs in the upper trapezius, confirmed via Travell and Simons' (1999) criteria (palpable taut band, spot tenderness, referred pain, and local twitch response);
* Chronic pain lasting 2-3 months; and
* Willingness to provide informed consent.

Exclusion Criteria:

* Fibromyalgia (per American College of Rheumatology criteria; Wolfe et al., 1990);
* Recent MTrP injections or physical therapy (within 1 year);
* Acute trauma or systemic conditions (e.g., inflammatory diseases); and
* Neurological deficits.
* Non-willingness to participation or showed non-cooperation.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 54 (Actual)
Dates: Start 2022-08-07 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Once a week for 3 weeks (baseline, week 1 and 2 post-intervention, and follow up at week 3 after one-week completion of intervention.
  Pain intensity was assessed using the visual analog scale (VAS), an imaginary line with either end marked with 0 or 10, indicating no pain or extremely unbearable pain, respectively.
Cervical range of motion | Once a week for 3 weeks (baseline, week 1 and 2 post-intervention, and follow up at week 3 after one-week completion of intervention.
  Cervical range of motion (ROM) was assessed with a universal goniometer for flexion, extension, right and left lateral flexion, and rotation.
Functional disability | Once a week for 3 weeks (baseline, week 1 and 2 post-intervention, and follow up at week 3 after one-week completion of intervention.
  Neck disability was quantified using the Neck Disability Index (NDI), a 10-item questionnaire with established reliability. The minimum and maximum scores are 0 and 50, indicating no disability to severe disability, respectively.
Upper trapezius muscle length | Once a week for 3 weeks (baseline, week 1 and 2 post-intervention, and follow-up at week 3 after one-week completion of intervention).
  Upper trapezius muscle length was measured using a vernier calliper with the participants seated in a standardized position. The distance between the mastoid process (posterior to the ear) and the acromioclavicular joint (distal end of the clavicle) was considered.

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University Hospital, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Khan N, Ghai T, Kashyap R, Bhat P, Ahmad F, Iqbal A, Alghadir T, Alghadir F, Anwer S, Alghadir AH. Comparative efficacy of myofascial release versus stretching combined with high-powered pulsed therapeutic ultrasound in amateur overhead athletes with active trapezius trigger point pain: a randomized clinical trial. BMC Sports Sci Med Rehabil. 2025 Dec 17. doi: 10.1186/s13102-025-01474-y. Online ahead of print. PMID 41402896
- See also: Controlled intervention to compare the efficacies of manual pressure release and the muscle energy technique for treating mechanical neck pain due to upper trapezius trigger points — https://doi.org/10.2147/JPR.S172711